CLINICAL TRIAL: NCT01138514
Title: A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study to Compare Perrigo Israel Pharmaceuticals, Ltd., Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel to a Comparator Clindamycin / Benzoyl Peroxide Topical Gel, and Both Active Treatments to a Vehicle Control in the Treatment of Acne Vulgaris
Brief Title: Clinical Study Between Two Clindamycin 1%/Benzoyl Peroxide 5% Topical Gels
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-716
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Benzoyl Peroxide; clindamycin phosphate benzoyl peroxide combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clindamycin 1%/Benzoyl Peroxide 5% (Active Comparator)
  Interventions: Drug: Clindamycin 1% / Benzoyl Peroxide 5% (Perrigo)
- Reference Product (Active Comparator)
  Interventions: Drug: Clindamycin 1% / Benzoyl Peroxide 5% (Benzaclin)
- Vehicle (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clindamycin 1% / Benzoyl Peroxide 5% (Perrigo) — Applied to the entire face twice daily for 10 weeks
  Arms: Clindamycin 1%/Benzoyl Peroxide 5%
Drug: Clindamycin 1% / Benzoyl Peroxide 5% (Benzaclin) — Applied to the entire face twice daily for 10 weeks
  Arms: Reference Product
Drug: Placebo — Placebo
  Arms: Vehicle

SUMMARY:
The purpose of this study is to compare the efficacy and safety profiles of Perrigo Israel Pharmaceuticals, Ltd. Clindamycin 1%/Benzoyl Peroxide 5% Topical Gel and Benzaclin® Topical Gel (Clindamycin- Benzoyl Peroxide Gel).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women, 12 to 65 years of age
* Willing to participate and sign provide written consent
* Moderate to severe acne

Exclusion Criteria:

* Pregnant or lactating women
* History of unresponsiveness or hypersensitivity to clindamycin, benzoyl peroxide or lincomycin
* Use of systemic, topical or facial products which may interfere with the study
* Participation in any clinical study in the 30 days prior to study entry
* Prolonged exposure to sunlight or excessive exposure to UV lights
* Chronic use of NSAIDS

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1555 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clindamycin 1%/Benzoyl Peroxide 5% | Reference Product | Vehicle
Started | 522 | 516 | 517
Completed | 474 | 463 | 424
Not Completed | 48 | 53 | 93

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clindamycin 1%/Benzoyl Peroxide 5% | Reference Product | Vehicle | Total
Number analyzed (Participants) | 522 | 516 | 517 | 1555
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.2 (7.6) | 20.1 (7.4) | 20.7 (8.1) | 20.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 284 | 282 | 279 | 845
  Male | 238 | 234 | 238 | 710
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 253 | 268 | 251 | 772
  Not Hispanic or Latino | 269 | 248 | 266 | 783
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3 | 6
  Asian | 11 | 10 | 10 | 31
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Black or African American | 90 | 80 | 98 | 268
  White | 308 | 310 | 296 | 914
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 110 | 114 | 109 | 333

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Inflammatory Lesions
Time Frame: 10 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percentage of lesion reduction
Arm/Group | Clindamycin 1%/Benzoyl Peroxide 5% | Reference Product | Vehicle
Number analyzed (Participants) | 430 | 419 | 427
percentage of lesion reduction | 79.87 (27.38) | 80.86 (24.65) | 45.60 (44.01)
Statistical Analysis 1: Comparison: Clindamycin 1%/Benzoyl Peroxide 5% vs Reference Product; Test type: Non-Inferiority or Equivalence — provides 85% power of success; p = 0.05, Fieller's method; equivalence ratio = 98.77, 90% CI 2-sided [95.2 to 102.5]

2. Primary Outcome: Percent Change From Baseline in Non-inflammatory Lesions
Time Frame: 10 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percentage of lesion reduction
Arm/Group | Clindamycin 1%/Benzoyl Peroxide 5% | Reference Product | Vehicle
Number analyzed (Participants) | 430 | 419 | 427
percentage of lesion reduction | 70.21 (30.48) | 70.02 (28.77) | 36.16 (48.15)
Statistical Analysis 1: Comparison: Clindamycin 1%/Benzoyl Peroxide 5% vs Reference Product; Test type: Non-Inferiority or Equivalence — provides 85% power of success; p = 0.05, Fieller's method; equivalence ratio = 100.27, 90% CI 2-sided [95.6 to 105.2]

3. Secondary Outcome: Number of Participant With Clinical Success on the Investigator's Global Assessment (IGA)
Description: Clinical success was defined as a score of clear (0) or almost clear (1) at Week 10.
Time Frame: 10 weeks
Population: per-protocol population
Measure: Number; unit: participants
Groups:
- Vehicle: Placebo
Arm/Group | Clindamycin 1%/Benzoyl Peroxide 5% | Reference Product | Vehicle
Number analyzed (Participants) | 430 | 419 | 427
participants | 247 | 234 | 79
Statistical Analysis 1: Comparison: Clindamycin 1%/Benzoyl Peroxide 5% vs Reference Product; Test type: Non-Inferiority or Equivalence — Clinical success was defined as a score of clear (0) or almost clear (1) on Investigator"s Global Assessment (IGA) at Visit 4/Week 10; p = 0.05, Wald's method Yates' continuity correct; equivalence difference = 1.6, 90% CI 2-sided [-4.2 to 7.4]

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Clindamycin 1%/Benzoyl Peroxide 5% | Reference Product | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/522 | 0/516 | 0/517
Other Adverse Events (participants affected / at risk) | 49/522 | 49/516 | 72/517
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clindamycin 1%/Benzoyl Peroxide 5% (N=522) | Reference Product (N=516) | Vehicle (N=517)
Application Site dryness (General disorders) | 32 (32) | 34 (34) | 6 (6)
Acne (Skin and subcutaneous tissue disorders) | 17 (17) | 16 (16) | 66 (66)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less